CLINICAL TRIAL: NCT01014624
Title: Recovery of Platelet Function Following Discontinuation of Prasugrel or Clopidogrel Maintenance Dosing in Aspirin-Treated Subjects With Stable Coronary Disease
Brief Title: Prasugrel/Clopidogrel Maintenance Dose Washout Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CS747S-B-U4001
Record Dates: First submitted 2009-11-16; First posted 2009-11-17 (Estimated); Results first posted 2011-09-09 (Estimated); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Coronary Artery Disease
Keywords: thienopyridine; pharmacologic action; prasugrel; clopidogrel
MeSH Terms: conditions — Coronary Artery Disease | interventions — Prasugrel Hydrochloride; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prasugrel (Experimental): Prasugrel 10mg administered for 7 days followed by a Washout Period up to 12 days.
  Interventions: Drug: Prasugrel
- Clopidogrel (Active Comparator): Clopidogrel 75mg administered for 7 days followed by a 12 day Washout Period up to 12 days.
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Prasugrel — Prasugrel 10mg tablet administered once daily for 7 days.
  After a 1-day to 14-day screening period, participants will receive active treatment with either prasugrel or clopidogrel for 7 days. If a participant has not missed more than 1 dose of study medication and is unable to attend Visit 3 (Washout Day 1) the day after the 7th day of study medication, the participant may take up to an additional 3 days of study medication and proceed to Visit 3 the day after the last dose. Active treatment will be followed by a 1-day to 12-day Washout Period depending on the time to reach both of the exit criteria.
  Other Names: Effient
  Arms: Prasugrel
Drug: Clopidogrel — Clopidogrel 75 mg tablet administered once daily for 7 days.
  After a 1-day to 14-day screening period, participants will receive active treatment with either prasugrel or clopidogrel for 7 days. If a participant has not missed more than 1 dose of study medication and is unable to attend Visit 3 (Washout Day 1) the day after the 7th day of study medication, the participant may take up to an additional 3 days of study medication and proceed to Visit 3 the day after the last dose. Active treatment will be followed by a 1-day to 12-day Washout Period depending on the time to reach both of the exit criteria.
  Other Names: Plavix
  Arms: Clopidogrel

SUMMARY:
The primary objective of the study is to describe the cumulative proportion of participants who return to baseline platelet P2Y12 receptor function over time (up to 12 days post last maintenance dose) following discontinuation of prasugrel 10 mg daily x 7 days assessed by Accumetrics VerifyNow P2Y12 reaction units (PRU) and described by Kaplan Meier curves. The primary analysis is descriptive and is intended to provide information relating to the return of baseline platelet function following discontinuation of maintenance therapy with either prasugrel or clopidogrel.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects >/= 18 years and <75 years of age
* Weight >/= 60 kg
* On aspirin therapy (81 mg to 325 mg daily) at the time of screening and able to maintain a consistent aspirin dosing regimen from the baseline visit through the final study visit
* Subjects who do not have contraindications for a thienopyridine (ie, prasugrel, clopidogrel or ticlopidine), and have a history of stable atherosclerosis represented by Coronary Artery disease, defined as any of the following:

  * chronic stable angina
  * Prior history of acute coronary syndrome (>/= 30 days before screening) including unstable angina or acute myocardial infarction (ST elevation Myocardial Infarction [STEMI] or non-ST elevation Myocardial Infarction [NSTEMI]), not currently prescribed or currently on thienopyridine therapy;
  * Previous coronary revascularization including percutaneous transluminal coronary angioplasty (PTCA), stent, or coronary artery bypass grafting (CABG) coronary artery disease (>/= 50% obstruction) in at least one coronary vessel after angiography
* Female subjects who meet one of the following:

  * Women of childbearing potential with a negative serum pregnancy test at screening who are not breast feeding, do not plan to become pregnant during the study, and agree to use an approved method of birth control during the study. Approved methods of birth control are oral, path, injectable or implantable hormonal contraception, intrauterine device, diaphragm plus spermicide, or female condom plus spermicide. Abstinence, partner's use of condoms, and partner's vasectomy are NOT acceptable methods of contraception.
  * Women who have been postmenopausal for at least 1 year or have had a hysterectomy, bilateral salpingo-oophorectomy, or tubal ligation at least 6 months prior to signing the informed consent form.
* Subjects with a competent mental condition to provide written informed consent before entering the study.

Exclusion Criteria:

* Any other formal indication for the use of a thienopyridine.
* Subjects with a history of refractory ventricular arrhythmias.
* Subjects with a history of an implantable defibrillator device.
* Subjects with a history or evidence of congestive heart failure (New York Heart Association [NYHA] Class III or above) within 6 months prior to screening.
* Subjects with significant hypertension (systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg) at either the time of screening or baseline assessment.
* Bleeding Risk Exclusion Criteria:

  * Any known contraindication to treatment with an anticoagulant or antiplatelet agent
  * Prior history or clinical suspicion of cerebral vascular malformations, intracranial tumor, transient ischemic attack (TIA), or stroke, or recent history (within 3 months) of head trauma
  * Prior history or presence of significant bleeding disorders (eg, hematemesis, melena, severe or recurrent epistaxis, hemoptysis, hematuria, or intraocular bleeding)
  * History (within the last 5 years) or presence of gastric ulcers. Previous history of duodenal ulcer is acceptable but must have been successfully surgically or medically treated with no further evidence of disease in the past 6 months (from screening).
  * Prior history of abnormal bleeding tendency (ie, prolonged bleeding on dental extraction, tonsillectomy, or previous surgical procedure)
  * Known prior history of thrombocytopenia (platelet count < 100,000/mm³) or thrombocytosis (platelet count > 500,000/mm³) or recent history (within six months) of hemoglobin < 10 mg/dL
  * Clinically significant out of range values for prothrombin time, activated partial thromboplastin time (aPTT), platelet count, or hemoglobin at screening, in the investigator's opinion
  * History of major surgery, severe trauma, fracture, or organ biopsy within 3 months prior to enrollment
* Prior/Concomitant Therapy Exclusion Criteria:

  * Subjects taking prasugrel, clopidogrel, ticlopidine, cilostazol, dipyridamole, warfarin, heparin, direct thrombin inhibitors, or glycoprotein IIB/IIIa inhibitors =10 days prior to screening or during study participation
  * The use (or planned use) of fibrinolytic agents within 30 days before screening or during study participation
  * Subjects receiving treatment with nonsteroidal anti-inflammatory drugs (NSAIDs) or cyclooxygenase-2 (COX-2) inhibitors exceeding 3 doses per week
  * Subjects receiving proton pump inhibitors (PPIs), eg, (lansoprazole, esomeprazole, omeprazole, pantoprazole, or rabeprazole) =10 days prior to screening or during study participation
* General Exclusion Criteria:

  * Investigator site personnel directly affiliated with the study or immediate family of investigator site personnel directly affiliated with the study. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted
  * Daiichi Sankyo or Eli Lilly employees
  * Currently enrolled in, or discontinued within the last 30 days prior to baseline from, a clinical study involving an off-label use of an investigational drug or device, or concurrently enrolled in a non-observational clinical study or any other type of medical research judged not to be scientifically or medically compatible with this study
  * Have previously completed or withdrawn from this study
  * Women who are known to be pregnant and/or who receive a positive serum pregnancy test result, who have given birth within the past 90 days, and/or who are breastfeeding
  * Results of clinical laboratory tests at the time of screening that are judged to be clinically significant for the subject, as determined by the investigator
  * Known allergies or intolerance to aspirin and/or thienopyridines (prasugrel, clopidogrel, or ticlopidine)
  * Evidence of significant active neuropsychiatric disease, alcohol abuse or drug abuse, in the investigator's opinion
  * Evidence of active hepatic disease, or any of the following; positive human immunodeficiency virus (HIV) antibodies, positive hepatitis C antibody, positive hepatitis B surface antigen; serum alanine transaminase (ALT), aspartate transaminase (AST), or gamma-glutamyltransferase (GGT) >/= 3 times the upper limit of normal (ULN) laboratory reference range; or bilirubin >/= 2 times the ULN of laboratory reference range at screening
  * Subjects who are unreliable and unwilling to make themselves available for the duration of the study and who will not abide by the research unit policy and procedure and study restrictions
* Subjects who have had an angiogram </= 7 days before randomization

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Scripps Clinic, La Jolla, California
  - University of Florida Health Science Center Shands Jacksonville, Jacksonville, Florida
  - Medpace Clinical Pharmacology Unit, Cincinnati, Ohio
  - Black Hills Clinical Research Center, Rapid City, South Dakota

REFERENCES:
- [Derived] Price MJ, Walder JS, Baker BA, Heiselman DE, Jakubowski JA, Logan DK, Winters KJ, Li W, Angiolillo DJ. Recovery of platelet function after discontinuation of prasugrel or clopidogrel maintenance dosing in aspirin-treated patients with stable coronary disease: the recovery trial. J Am Coll Cardiol. 2012 Jun 19;59(25):2338-43. doi: 10.1016/j.jacc.2012.02.042. PMID 22698488

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 4 sites in the US from 23 February 2010 to 24 May 2010 and 56 participants were randomized into the study. The study population consisted of male and female aspirin-treated participants with stable coronary artery disease, 18 to 75 years of age.
Pre-assignment Details: The Overall Study Period included a 1-day to 14-day Screening Period, a 7-day Active Treatment Period, and a Washout Period of up to 12 days. Following the 1-day to 14-day Screening Period, eligible participants were randomized in a 1:1 ratio to either prasugrel or clopidogrel at Visit 2 (the first day of the Active Treatment Period).
Groups:
- Prasugrel: Prasugrel 10mg tablet administered once daily for 7 days followed by a Washout Period up to 12 days.
- Clopidogrel: Clopidogrel 75 mg tablet administered once daily for 7 days followed by Washout Period up to 12 days.
Period: Overall Study
Arm/Group | Prasugrel | Clopidogrel
Started | 29 | 27
Completed | 27 | 26
Not Completed | 2 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prasugrel | Clopidogrel | Total
Number analyzed (Participants) | 29 | 27 | 56
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.5 (8.45) [0 to 0] | 62.3 (8.10) [0 to 0] | 59.80 (8.56) [0 to 0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 25 | 20 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 28 | 27 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 22 | 22 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
weight [Mean (Standard Deviation); unit: kg] | 97.3 (15.13) [0 to 0] | 90.8 (14.41) [0 to 0] | 94.1 (15.02) [0 to 0]
Height [Mean (Standard Deviation); unit: cm] | 174.1 (8.20) [0 to 0] | 173.5 (9.00) [0 to 0] | 173.8 (8.52) [0 to 0]
Ethnicity [Number; unit: participants]
  Hispanic or Latino | 1 (0) [0 to 0] | 0 (0) [0 to 0] | 1 (0) [0 to 0]
  Non Hispanic or Latino | 28 (0) [0 to 0] | 27 (0) [0 to 0] | 55 (0) [0 to 0]
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 32.0 (4.07) [0 to 0] | 30.3 (5.34) [0 to 0] | 31.2 (4.76) [0 to 0]
Smoking Status [Number; unit: participants]
  Never smoked | 7 (0) [0 to 0] | 10 (0) [0 to 0] | 17 (0) [0 to 0]
  Currently Smoke | 10 (0) [0 to 0] | 6 (0) [0 to 0] | 16 (0) [0 to 0]
  Formerly Smoked | 12 (0) [0 to 0] | 11 (0) [0 to 0] | 23 (0) [0 to 0]
Alcohol Use [Number; unit: participants]
  Never used alcohol | 3 (0) [0 to 0] | 5 (0) [0 to 0] | 8 (0) [0 to 0]
  Currently use alcohol | 19 (0) [0 to 0] | 18 (0) [0 to 0] | 37 (0) [0 to 0]
  Formerly used alcohol | 7 (0) [0 to 0] | 4 (0) [0 to 0] | 11 (0) [0 to 0]
Diabetes status [Number; unit: participants]
  Does not have diabetes | 18 (0) [0 to 0] | 16 (0) [0 to 0] | 34 (0) [0 to 0]
  Has diabetes | 11 (0) [0 to 0] | 11 (0) [0 to 0] | 22 (0) [0 to 0]

OUTCOME MEASURES:

1. Primary Outcome: The Time to Return to Baseline Platelet Function as Assessed by P2Y12 Reaction Units (PRU) Using the Accumetrics VerifyNOW P2Y12 Device Based on the Primary Definition of Return to Baseline
Description: On the first day of the Washout Period (Visit 3), the blood draw for platelet function testing was obtained 24 hours (+/- 6 hours) after the last dose of study medication. Following Visit 3, platelet function testing was performed during each visit of the Washout Period until the participant met the following exit criteria: (Baseline PRU-PRU) less than or equal to 60 units and (Baseline PRU-PRU)/(Baseline PRU) less than or equal to 20%. The results are expressed as cumulative percentage of participants.
Time Frame: up to 12 days after last dose
Population: Participants in Primary Population defined as Baseline PRU-PRU less than or equal to 60 units (R-to-B). Primary Population included participants who entered Washout Period and had platelet function data at both baseline and Washout Period Day 1.
Measure: Number; unit: cumulative percentage of participants
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 28 | 26
cumulative percentage of participants
  return to baseline PRU by washout day 1 | 0 | 30.8
  return to baseline PRU by washout day 3 | 3.6 | 53.9
  return to baseline PRU by washout day 5 | 37.0 | 84.6
  return to baseline PRU by washout day 6 | 62.9 | 96.2
  return to baseline PRU by washout day 7 | 77.8 | 96.2
  return to baseline PRU by washout day 9 | 100.0 | 100.0

2. Primary Outcome: The Time to Return to Baseline Platelet Function as Assessed by P2Y12 Reaction Units (PRU) Using the Accumetrics VerifyNOW P2Y12 Device Based on the Secondary Definition of Return to Baseline
Description: On the first day of the Washout Period (visit 3), the blood draw for platelet function testing was obtained 24 hours (+/- 6 hours) after the last dose of study medication. Following Visit 3, platelet function testing was performed during each visit of the Washout Period until the participant met the following exit criteria: (Baseline PRU-PRU) less than or equal to 60 units and (Baseline PRU-PRU)/(Baseline PRU) less than or equal to 20%.
Time Frame: up to 12 days after last dose
Population: Participants in Primary Population using secondary definition of return to baseline. Primary Population included participants who entered the Washout Period and had platelet function data at both baseline and Washout Period Day 1. Secondary definition of return to baseline was (Baseline PRU-PRU)/Baseline PRU less than or equal to 20%.
Measure: Number; unit: cumulative percentage of participants
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 28 | 26
cumulative percentage of participants
  returned to baseline PRU by washout day 1 | 0.0 | 30.8
  returned to baseline PRU by washout day 3 | 0.0 | 53.9
  returned to baseline PRU by washout day 5 | 37.0 | 80.8
  returned to baseline PRU by washout day 6 | 55.6 | 88.5
  returned to baseline PRU by washout day 7 | 77.8 | 96.2
  returned to baseline PRU by washout day 9 | 100.0 | 100.0

3. Secondary Outcome: Day at Which 50%, 75%, and 90% of Participants Returned to Baseline Platelet Function Based on Primary Definition of Return to Baseline Using the Primary Population
Description: On the first day of the Washout Period (Visit 3), the blood draw for platelet function testing was obtained 24 hours (+/-6 hours) after the last dose of study medication. Following Visit 3, platelet function testing was performed during each visit of the Washout Period until the participants met the following exit criteria: (Baseline PRU-PRU) less than or equal to 60 units and (Baseline PRU-PRU)/Baseline PRU less than or equal to 20%.
Time Frame: up to 12 days after last dose
Population: Participants in Primary Population using primary definition of return to baseline. Primary population included participants who entered the Washout Period and had platelet function data at both baseline and Washout Period Day 1. Primary definition of return to baseline was (Baseline PRU-PRU) less than or equal to 60 units.
Measure: Number; unit: days
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 28 | 26
days
  Washout day 50% returned to baseline PRU | 6 | 3
  Washout day 75% returned to baseline PRU | 7 | 5
  Washout day 90% returned to baseline PRU | 9 | 6

4. Secondary Outcome: Day at Which 50%, 75%, and 90% of Participants Returned to Baseline Platelet Function Based on Secondary Definition of Return to Baseline Using the Primary Population
Description: On the first day of the Washout Period (Visit 3), the blood draw for platelet function testing was obtained 24 hours (+/-6 hours) after the last dose of study medication. Following Visit 3, platelet function testing was performed during each visit of the Washout Period until the participant met the following exit criteria: (Baseline PRU-PRU) less than or equal to 60 units and (Baseline PRU-PRU)/Baseline PRU less than or equal to 20%.
Time Frame: up to 12 days after last dose
Population: Participants in Primary Population using secondary definition of return to baseline. Primary Population included participants who entered Washout Period and had platelet function data at both baseline and Washout Period Day 1. Secondary definition of return to baseline was (Baseline PRU-PRU)/Baseline PRU less than or equal to 20%.
Measure: Number; unit: days
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 28 | 26
days
  Washout day 50% returned to baseline PRU | 6 | 3
  Washout day 75% returned to baseline PRU | 7 | 5
  Washout day 90% returned to baseline PRU | 9 | 7

5. Secondary Outcome: Day at Which 50%, 75%, and 90% of Participants Returned to Baseline Platelet Function Based on the Primary Definition of Return to Baseline Using the Responder Population
Description: as for outcome 4
Time Frame: up to 12 days after last dose
Population: Participants in Responder Population using primary definition of R-to-B. Primary Population included participants who entered Washout Period and had platelet function data at baseline and Washout Day 1. Responder Population was Primary Population excluding poor pharmacodynamic responders. Primary definition of R-to-B was (Baseline PRU-PRU) less than or equal to 60 units.
Measure: Number; unit: days
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 28 | 15
days
  Washout day 50% returned to baseline PRU | 6 | 5
  Washout day 75% returned to baseline PRU | 7 | 5
  Washout day 90% returned to baseline PRU | 9 | 6

6. Secondary Outcome: Day at Which 50%, 75%, and 90% of Participants Returned to Baseline Platelet Function Based on the Secondary Definition of Return to Baseline Using the Responder Population
Description: On the first day of the Washout Period (Visit 3), the blood draw for platelet function testing was obtained 24 hour (+/- 6 hours) after the last dose of study medication. Following Visit 3, platelet function testing was performed during each visit of the Washout Period until the participant met the following exit criteria: (Baseline PRU-PRU) less than or equal to 60 units and (Baseline PRU-PRU)/(Baseline PRU) less than or equal to (<=) 20%.
Time Frame: up to 12 days after the last dose
Population: Participants in Responder Population using secondary definition of R-to-B. Primary Population included participants who entered Washout Period and had platelet function data at both baseline and Washout Period Day 1. Responder Population was Primary Population excluding poor pharmacodynamic responders. Secondary definition of R-to-B was (Baseline PRU-PRU)/ (Baseline PRU) <= 20%.
Measure: Number; unit: days
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 28 | 15
days
  Washout day 50% returned to baseline PRU | 6 | 5
  Washout day 75% returned to baseline PRU | 7 | 6
  Washout day 90% returned to baseline PRU | 9 | 7

7. Secondary Outcome: Percentage of Inhibition of Platelet Aggregation on Washout Day 1
Description: Inhibition of platelet aggregation was assessed by Accumetrics VerifyNow® P2Y12 reaction units (PRU). On the first day of the Washout Period (Visit 3), the blood draw for platelet function testing was obtained 24 hour (+/- 6 hours) after the last dose of study medication. Following Visit 3, platelet function testing was performed during each visit of the Washout Period until the participant met the following exit criteria: (Baseline PRU-PRU) less than or equal to 60 units and (Baseline PRU-PRU)/(Baseline PRU) less than or equal to 20%.
Time Frame: Washout Day 1
Population: Participants in the Primary Population. The Primary Population included participants who entered the Washout Period and had platelet function testing data at both baseline (Visit 2) and Washout Period Day 1 (Visit 3).
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 28 | 26
percentage | 72.3 (11.78) | 35.4 (23.35)

8. Secondary Outcome: Time to Return to Baseline PRU for the Primary Population Using the Primary Definition of Return to Baseline in Relation to the Inhibition of Platelet Aggregation 24 Hours Following the Last Maintenance Dose
Description: Time to return to baseline PRU (<= 60 units of baseline) dependent upon baseline PRU and platelet % inhibition on Washout Period Day 1 but independent of treatment. The following regression model was derived for predicting number of days to return to baseline PRU where PI(1) represents platelet percentage inhibition on Washout Day 1. Number days to return to baseline PRU derived from: Number days to return to baseline PRU=-3.350+0.079*PI(1)+0.014*baseline PRU. The predicted number of days to return to baseline based on device-derived platelet percentage inhibition is reported for each treatment group.
Time Frame: up to 12 days after the last dose
Population: Participants in the Primary Population. The Primary Population included participants who entered the Washout Period and had platelet function testing data at both baseline (Visit 2) and Washout Period Day 1 (Visit 3). The primary definition of return to baseline was (Baseline PRU-PRU) less than or equal to 60 units.
Measure: Number; unit: days
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 28 | 26
days | 6.2 | 3.7

ADVERSE EVENTS:
Time Frame: Beginning with screening, adverse events (AEs) were assessed at every visit. All AEs occuring after participant signed informed consent and up to 14 days after last dose of study drug were recorded
Arm/Group | Prasugrel | Clopidogrel
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/27
Other Adverse Events (participants affected / at risk) | 12/29 | 9/27
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prasugrel (N=29) | Clopidogrel (N=27)
eyelid oedema (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Adominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
viral infection (Infections and infestations) | 1 (1) | 0 (0)
diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
dizziness (Nervous system disorders) | 1 (1) | 0 (0)
headache (Nervous system disorders) | 1 (1) | 0 (0)
insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
increased tendency to bruise (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Adominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No